CLINICAL TRIAL: NCT06594341
Title: Operational Pilot Study for Treatment of Acute Malnutrition with Simplified Approaches in Mali
Brief Title: Optimization of the Simplified Protocol in Mali: a Cluster Randomised Pragmatic Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: International Rescue Committee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: H.1.00.025
Record Dates: First submitted 2023-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Acute Malnutrition in Infancy; Acute Malnutrition in Childhood; Acute Malnutrition, Severe
MeSH Terms: conditions — Severe Acute Malnutrition

STUDY DESIGN:
Intervention Model Description: A total of 39 health areas including 39 health centers and 52 secondary sites will be be randomised into : 1) providing simplified treatment as per on-going routine protocol, 2) providing simplified treatment with a reduced visit frequency for children in the moderate phase, 3) providing simplified treatment without a transition period for children admitted with severe malnutrition when they progress to moderate phase and 4) providing simplified treatment with a reduced visit frequency for children in the moderate phase and without a transition phase for children admitted with severe malnutrition when they porgress to modera phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Simplified treatment (Active Comparator): Children will be treated with a simplified protocol prescribing 2 sachets of RUTF to children admitted with a MUAC<115mm or edema and 1 sachet to children with MUAC 115-124mm. Children admitted with a MUAC<115mm or edema will be transitioned to receive 1 sachet of RUTF once they have reached a MUAC>=115mm for 2 consecutive visits. Visit frequency will be weekly for all children regardless of severity or phase.
  Interventions: Procedure: Simplified treatment
- Simplified treatment with a reduced visit frequency (Experimental): Children will be treated with a simplified protocol prescribing 2 sachets of RUTF to children admitted with a MUAC<115mm or edema and 1 sachet to children with MUAC 115-124mm. Children admitted with a MUAC<115mm or edema will be transitioned to receive 1 sachet of RUTF once they have reached a MUAC>=115mm for 2 consecutive visits. Visit frequency will be weekly for children in the "severe phase" and fortnightly for children in the "moderate" phase.
  Interventions: Procedure: Visit frequency; Procedure: Simplified treatment
- Simplified treatment without transition period (Experimental): Children will be treated with a simplified protocol prescribing 2 sachets of RUTF to children admitted with a MUAC<115mm or edema and 1 sachet to children with MUAC 115-124mm. Children admitted with a MUAC<115mm or edema will be transitioned to receive 1 sachet of RUTF immediately when they have reach a MUAC>=115mm. Visit frequency will be weekly for all children regarless of severity or phase.
  Interventions: Dietary Supplement: Suppression of the transition period; Procedure: Simplified treatment
- Simplified treatment with a reduced visit frequency and without a transition period (Experimental): Children will be treated with a simplified protocol prescribing 2 sachets of RUTF to children admitted with a MUAC<115mm or edema and 1 sachet to children with MUAC 115-124mm. Children admitted with a MUAC<115mm or edema will be transitioned to receive 1 sachet of RUTF immediately once reach a MUAC>=115mm . Visit frequency will be weekly for children in the "severe phase" and fortnightly for children in the "moderate" phase.
  Interventions: Procedure: Visit frequency; Dietary Supplement: Suppression of the transition period; Procedure: Simplified treatment

INTERVENTIONS:
Procedure: Visit frequency — Fortnightly visit frequency for moderate phase
  Nutritional supplement: 1 daily sachet of RUTF as soon as a child admitted with MUAC<115mm or edema reaches a MUAC=>115mm or absence of edema.
  Arms: Simplified treatment with a reduced visit frequency; Simplified treatment with a reduced visit frequency and without a transition period
Dietary Supplement: Suppression of the transition period — Transitioning children admitted with MUAC<115mm or edema to receiving 1 daily sachet of RUTF as soon as they reach a MUAC=>115mm and absence of edema
  Arms: Simplified treatment with a reduced visit frequency and without a transition period; Simplified treatment without transition period
Procedure: Simplified treatment — Admitting children with MUAC<125mm or edema to treatment prescribing 2 daily sachets for children with MUAC<115mm or edema and 1 daily sachet for children with MUAC 115mm to 124mm. Treatment visits are done on a weekly basis and children with MUAC<115mm are transitioned to receiving 1 daily sachet of RUTF once they reach a MUAC=>115mm for 2 consecutive measurements. Treatment is continued until recovery defined as a MUAC=>125mm for 2 consecutive weeks.

SUMMARY:
Acute malnutrition is a condition that affects more than 45 million children under the age of five at any time and requires specific treatment to ensure patient survival. Most patients can be managed as outpatients with regular monitoring to ensure the correct evolution of nutritional status. With adequate treatment the cure rate of children is high and few patients die.

At the same time, despite the existence of an effective protocol for treating malnutrition at the level of health structures, current strategies do not make it possible to reach all malnourished children. On the global level, it is estimated that only 20% of children in need of treatment actually receive it.

In Mali, in order to improve coverage and quality of malnutrition treatment in children under five, an operational pilot on simplified approaches to treatment was launched in 2018 and has been on-going since in the health district of Nara.

The three simplifications being implemented include:

1. treatment of acute malnutrition using a simplified protocol and an optimized dosage for both SAM and MAM at the health facility;
2. treatment at community level by community health volunteers (CHWs) of acute malnutrition using the same simplified protocol and an optimized dosage;
3. scale up of the use of MUAC bands by caregivers to identify and monitor their children's nutritional status, also known as family MUAC.

This approach has been implemented throughout the Health District (HD) of Nara in the Koulikoro Region comprising 39 health centers, 52 ASC functional sites and 11 rural maternities. The simplified treatment of children is done by regular MoH staff with IRC providing technical support and a reinforced monitoring and evaluation of treatment outcomes.

In order to strengthen the evidence on the effects of simplified approaches on the treatment of acute malnutrition, IRC is collecting regular patient data to monitor the treatment outcomes of the patients. This data is used to analyze the recovery rate of children, the length of stay in treatment, the mean weight gain velocity etc. Rigorous programmatic data on such large scale operational pilots is crucial for documenting the real life performance of the simplified approaches and provide evidence on the potential of this approach for scale up. In 2022, IRC published an article on the programmatic results of the pilot showing very high recovery among children treated with the simplified protocol.

However, while the simplified treatment seems to be working well in this contexts, both health care workers administering treatment as well as caregivers of treated children have suggested further simplifications to the protocol.

In order to document potential impact of such changes on the treatment effectiveness, we propose to make these changes in a sub-set of health areas currently implementing the simplified protocol and run this study as a pragmatic cluster randomised trial. The changes to be tested in the first phase include 1) further simplifying the transition period observed among children admitted with severe malnutrition before they start receiving a lower dose of treatment and 2) spacing out treatment visits from weekly to fortnightly.

Other small adjustments to the treatment protocol could be tested in the future in a similar way.

ELIGIBILITY:
Inclusion Criteria:

* MUAC<125mm or edema at admission to treatment
* treated with the simplified protocol in one of the treatment facilities participating in study

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6249 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2024-02-10 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
recovery | from admission to maximum 16 weeks post-admission
  percent of children recovered (defined as MUAC>=125mm for 2 consecutive measures)

SECONDARY OUTCOMES:
defaulting | from admission to discharge at maximum 16 weeks post-admission
  percent of children who end up missing 2 or more treatment visits and being declared defaulted
diseased | from admission to discharge at maximum 16 weeks post-admission
  percent of children who die during treatment
length of stay in treatment | from admission to discharge (recovered, non-recovered, defaulted or died) at maximum 16 weeks post-admission
  average number of days from admission to discharge from treatment
RUTF consumed | from admission to discharge (recovered, non-recovered, defaulted, died) at maximum 16 weeks post-admission
  average number of RUTF sachets consumed from admission to discharge
non-recovery | from admission to discharge at maximum 16 weeks post-admission
  percent of children not having recovered within 16 weeks of treatment

OTHER OUTCOMES:
cost of treatment | from admission to discharge (recovered, non-recovered, defaulted, died) from treatment at maximum 16 weeks after admission.
  including cost for the implementing partner, cost of products, cost to health system and cost to caregivers

CONTACTS AND LOCATIONS:
Locations (1):
- Nara district, Nara, Koulikoro, Mali

IPD SHARING:
Plan to Share IPD: Yes
We plan to make the de-identified data available for other researchers upon request and also publish the de-identified data sets that underlie the results of any scientific publications.
Supporting Information: SAP, Analytic Code
Time Frame: upon publication of any results from the study
Access Criteria: analysis plan describing the justification of the study, the research question, the hypothesis and objectives.
URL: https://zenodo.org/records/7343363